CLINICAL TRIAL: NCT07396584
Title: A Phase I/Ⅱa Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of HMPL-A580 in Participants With Advanced or Metastatic Solid Tumors
Brief Title: A Phase I/Ⅱa Study of HMPL-A580 in Participants With Advanced or Metastatic Solid Tumor
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-580-GLOB1
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A(Phase I) Dose Escalation (Experimental)
  Interventions: Drug: HMPL-A580
- Part B(Phase IIa) Dose Expansion/Dose Optimization (Experimental)
  Interventions: Drug: HMPL-A580

INTERVENTIONS:
Drug: HMPL-A580 — Part A(Phase I) Dose Escalation Enrolled participants will receive HMPL-A580 treatment in a dose escalation setting initially at 6 predefined dose levels.
  Arms: Part A(Phase I) Dose Escalation
Drug: HMPL-A580 — Part B(Phase IIa) Dose Expansion/Dose Optimization Evaluate the safety and preliminary anti-tumor activity of HMPL-A580 in selected solid tumors.
  Arms: Part B(Phase IIa) Dose Expansion/Dose Optimization

SUMMARY:
This is a first-in-human, multicenter, open-label, phase I/Ⅱa clinical study of HMPL-A580 in participants with unresectable, advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
To evaluate the safety, tolerability, and determine the maximum tolerated dose (MTD) and/or recommended dose(s) for expansion (RDE) of HMPL-A580 in solid tumors.

To characterize the safety, tolerability, and preliminary efficacy of HMPL-A580 at RDE(s) to determine recommended dose(s) for phase 2 dose (RP2D) or phase 3 dose (RP3D) in participants with selected solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Understood this study and are able to voluntarily sign the informed consent form (ICF);
2. Male or Female, Age ≥ 18 years;
3. Histological confirmed, unresectable, advanced or metastatic solid tumor
4. Participants must have at least one measurable lesion per RECIST v1.1
5. Life expectancy ≥ 12 weeks
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1

Exclusion Criteria:

1. An established diagnosis of type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus
2. Use strong inhibitors of cytochrome P450 3A4 enzyme (CYP3A4), and inhibitors of P-glycoprotein (P-gp) and breast cancer resistance protein (BCRP) within 5 elimination half-lives or 2 weeks (whichever is longer) before the first dose of study drug
3. Major surgery within 28 days prior to the first dose of study drug
4. Active infection requiring systemic treatment
5. Participant has received a live within 3 months before study enrollment
6. History of inflammatory gastrointestinal diseases
7. Known hypersensitivity to any component of HMPL-A580
8. Pregnant (positive pregnancy test) or lactating;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or recommended dose(s) for expansion(RDE) | Approximately 12 months
  To evaluate the safety, tolerability, and MTD) and/or RDE of HMPL-A580 in solid tumors
Overview of Treatment-emergent Adverse Events (TEAEs) | Approximately 12 months
  To characterize the safety of HMPL-A580 at RDE(s)
Objective Response Rate (ORR) | At least 8 weeks post dose of first participant up to approximately 24 months
  To characterize the tolerability, and preliminary efficacy of HMPL-A580 at RDE(s)
Recommended doses for phase II or III studies (RP2D or RP3D) of HMPL-A580 | Approximately 12 months
  To characterize the safety, tolerability, and preliminary efficacy of HMPL-A580 at RDE(s) to determine recommended dose(s) for phase 2 dose (RP2D) or phase 3 dose (RP3D) in participants with selected solid tumors.

SECONDARY OUTCOMES:
disease control rate (DCR) | Approximately 2 years
  To assess the preliminary efficacy of HMPL-A580 in solid tumors
progression-free survival (PFS) | Approximately 2 years
  To assess the preliminary antitumor activity of HMPL-A580 in selected solid tumors

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Hunan Cancer Hospital, Changsha
  - Guangxi Medical University Cancer Hospital, Nanning
  - Shanghai East Hospital, Shanghai
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Henan Cancer Hospital, Zhengzhou